CLINICAL TRIAL: NCT03765073
Title: A PHASE 1/2, RANDOMIZED, PLACEBO-CONTROLLED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MULTIVALENT GROUP B STREPTOCOCCUS VACCINE IN HEALTHY NONPREGNANT WOMEN AND PREGNANT WOMEN 18 TO 40 YEARS OF AGE AND THEIR INFANTS
Brief Title: Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of A Multivalent Group B Streptococcus Vaccine In Healthy Nonpregnant Women And Pregnant Women And Their Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: C1091002; 2020-005074-96 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Group B Streptococcus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is an observer-blinded study. Study staff dispensing and administering the vaccine will be unblinded, but all other study personnel, including the principal investigator, and the participant, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Stage 1 - Highest dose formulation a (Experimental): Multivalent group B streptococcus vaccine - Stage 1 Nonpregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 1 - Highest dose formulation b (Experimental): Multivalent group B streptococcus vaccine - Stage 1 Nonpregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Lowest dose formulation a (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Lowest dose formulation b (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Middle dose formulation a (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Middle dose formulation b (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Highest dose formulation a (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 2 - Highest dose formulation b (Experimental): Multivalent group B streptococcus vaccine - Stage 2 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 3 - Selected dose and formulation (Experimental): Multivalent group B streptococcus vaccine - Stage 3 Pregnant women
  Interventions: Biological: Multivalent Group B streptococcus vaccine
- Stage 1 Placebo (Placebo Comparator): Saline control
  Interventions: Biological: Placebo
- Stage 2 Placebo (Placebo Comparator): Saline control
  Interventions: Biological: Placebo
- Stage 3 Placebo (Placebo Comparator): Saline control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Multivalent Group B streptococcus vaccine — Various formulations at three dose levels
  Arms: Stage 1 - Highest dose formulation a; Stage 1 - Highest dose formulation b; Stage 2 - Highest dose formulation a; Stage 2 - Highest dose formulation b; Stage 2 - Lowest dose formulation a; Stage 2 - Lowest dose formulation b; Stage 2 - Middle dose formulation a; Stage 2 - Middle dose formulation b; Stage 3 - Selected dose and formulation
Biological: Placebo — Saline control
  Arms: Stage 1 Placebo; Stage 2 Placebo; Stage 3 Placebo

SUMMARY:
Phase 1/2, randomized, placebo-controlled, observer-blinded study will evaluate the safety, tolerability and immunogenicity of the investigational multivalent group B streptococcus vaccine administered at one dose level (various formulations) in healthy nonpregnant women (various formulations at one dose level), and then in healthy pregnant women (various formulations at three dose levels), and finally in healthy pregnant women at a selected dose level/formulation.

ELIGIBILITY:
Inclusion Criteria Stage 1 Nonpregnant Women:

* Healthy nonpregnant females 18 to 40 years of age at enrollment who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
* Negative urine pregnancy test at Visit 1 (prior to vaccination).
* Documented negative HIV, hepatitis C virus (HCV), and acute or chronic hepatitis B virus (HBV) infection at screening.

Inclusion Criteria Stage 1 Booster Vaccination:

* Participant must have received investigational product at Visit 1.
* Healthy nonpregnant female determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for booster vaccination and received investigational product at Visit 1.
* Negative urine pregnancy test at Visit 6 (prior to vaccination).
* Documented negative HIV, hepatitis C virus (HCV), and acute or chronic hepatitis B virus (HBV) infection at screening.

Inclusion Criteria Stage 2 and 3 Maternal Participants:

* Healthy females >=18 and <=40 years of age who are >=27 0/7 (Stage 2) or >=24 0/7 (Stage 3) to <=35 6/7 weeks' gestation on the day of planned vaccination, with an uncomplicated, singleton pregnancy, and at no increased risk for complications and no significant fetal abnormalities observed on ultrasound performed at any time prior to study entry and/or at the screening visit.
* Documented negative HIV antibody, HBV surface antigen, HCV antibody, and syphilis tests at screening.

Inclusion Criteria Stage 2 and 3 Infant Participants:

Evidence of a signed and dated ICD signed by the parent(s). Parent(s) willing and able to comply with scheduled visits, investigational plan, laboratory tests, and other study procedures.

Exclusion Criteria Stage 1 Nonpregnant Women:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product or any diphtheria toxoid-containing or CRM197 containing vaccine.
* History of microbiologically proven invasive disease caused by GBS (S agalactiae).
* Previous vaccination with any licensed or investigational GBS vaccine (other than GBS6 received as a primary vaccination at Visit 1), or planned receipt during the participant's participation in the study (through the last blood draw).

Exclusion criteria Stage 2 and 3 Maternal Participants:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product or any diphtheria toxoid-containing or CRM197 containing vaccine.
* History of microbiologically proven invasive disease caused by GBS (S agalactiae).
* Previous vaccination with any licensed or investigational group B streptococcus vaccine, or planned receipt during the participant's participation in the study (through the last blood draw).
* Prepregnancy body mass index (BMI) of ≥40 kg/m2. If prepregnancy BMI is not available, the BMI at the time of the first obstetric visit during the current pregnancy may be used.
* A prior history of or current pregnancy complications or abnormalities that will increase the risk associated with the participant's participation.
* Major illness of the mother or conditions of the fetus that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in, and completion of, the study or could preclude the evaluation of the participant's response.

Exclusion criteria Stage 2 and 3 Infant Participants:

Infant who is a direct descendant (eg, child or grandchild) of the study personnel.

Ages: 0 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1208 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (26):
  - Velocity Clinical Research, Mobile, Alabama
  - Velocity Clinical Research, Phoenix, Phoenix, Arizona
  - Chemidox Clinical Trials Inc., Lancaster, California
  - Chemidox Clinical Trials Inc, Lancaster, California
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Clinical Research Prime Rexburg, Rexburg, Idaho
  - Lakeview Regional Medical Center, Covington, Louisiana
  - MedPharmics, Covington, Louisiana
  - St. Tammany Parish Hospital, Covington, Louisiana
  - North Oaks Medical Center, Hammond, Louisiana
  - North Oaks Obstetrics & Gynecology, Hammond, Louisiana
  - Velocity Clinical Research, Slidell, Louisiana
  - Boeson Research, Missoula, Montana
  - Community Hospital, Missoula, Montana
  - The Birth Center, Missoula, Montana
  - Meridian Clinical Research, Hastings, Nebraska
  - Frontier Pediatric Care (Follow-Up Visits for Infant Participants), Lincoln, Nebraska
  - Bryan Women's Care Physicians (Maternal Visits & Obstetric Exams), Lincoln, Nebraska
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Lowcountry Women's Specialists, Summerville, South Carolina
  - Summerville Medical Center, Summerville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Sentara Leigh Hospital, Norfolk, Virginia
  - The Group for Women, Norfolk, Virginia
  - Tidewater Physicians for Women, Norfolk, Virginia
- South Africa (8):
  - Wits Reproductive Health and HIV Institute, Johannesburg, Gauteng
  - Respiratory and Meningeal Pathogens Research Unit (RMPRU), Soweto, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
  - Empilweni Services and Research Unit (ESRU), Coronationville, Johannesburg
  - Khayelitsha District Hospital (KDH), Khayelitsha, Western Cape
  - Michael Mapongwana Community Health Centre, Khayelitsha, Western Cape
  - Site B, Khayelitsha, Western Cape
  - FAMCRU, Parow Valley, Western Cape
- St George's University Hospitals NHS Foundation Trust, London, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cutland CL, Sawry S, Fairlie L, Barnabas S, Frajzyngier V, Roux JL, Izu A, Kekane-Mochwari KE, Vika C, De Jager J, Munson S, Jongihlati B, Stark JH, Absalon J. Obstetric and neonatal outcomes in South Africa. Vaccine. 2024 Feb 27;42(6):1352-1362. doi: 10.1016/j.vaccine.2024.01.054. Epub 2024 Feb 3. PMID 38310014
- [Derived] Madhi SA, Anderson AS, Absalon J, Radley D, Simon R, Jongihlati B, Strehlau R, van Niekerk AM, Izu A, Naidoo N, Kwatra G, Ramsamy Y, Said M, Jones S, Jose L, Fairlie L, Barnabas SL, Newton R, Munson S, Jefferies Z, Pavliakova D, Silmon de Monerri NC, Gomme E, Perez JL, Scott DA, Gruber WC, Jansen KU. Potential for Maternally Administered Vaccine for Infant Group B Streptococcus. N Engl J Med. 2023 Jul 20;389(3):215-227. doi: 10.1056/NEJMoa2116045. PMID 37467497
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1091002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy non-pregnant participants, pregnant maternal participants between 18 to 40 years of age and infants who were born to these maternal participants were enrolled in this study. This study conducted in three stages and participants were enrolled to Stage 1, 2 and 3 separately.
Pre-assignment Details: A total of 66 nonpregnant women and 576 maternal participants and their 566 infants were enrolled in this study. Infants were not randomized and vaccinated in this study but summarized according to the vaccine group their mothers were randomized to. Vaccination was administered preferably to the nondominant arm of the participants.
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 microgram of Group B Streptococcus 6-valent (GBS6) vaccine with aluminium phosphate, intramuscularly, preferably in nondominant arm on Day 1.
- Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly, preferably in nondominant arm on Day 1.
- Stage 1: Placebo (Nonpregnant): Non pregnant participants were randomized to receive placebo (saline control) intramuscularly, preferably in nondominant arm on Day 1.
- Stage 2: GBS6 5 mcg With AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 5 μg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 5 mcg Without AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 5 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg With AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 10 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg Without AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 10 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg With AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg Without AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: Placebo (Maternal); Stage 3: Placebo (Maternal): Maternal participants were randomized to receive placebo (saline control) intramuscularly on Day 1.
- Stage 2: GBS6 5 mcg With AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 5 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 5 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 5 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg With AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 10 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 10 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg With AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg Without AlPO4 (Infant); Stage 3: GBS6 20 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: Placebo (Infant): Infant participants born to the maternal participants randomized to receive placebo (saline control) intramuscularly on Day 1.
- Stage 3: GBS6 20 mcg Without AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AIPO4, intramuscularly on Day 1.
- Stage 3: Placebo (Infant): Infant participants were randomized to receive placebo (saline control) intramuscularly on Day 1.
Period: Stage 1
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Started | 22 | 22 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Booster Vaccination | 11 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 21 | 21 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by participant | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Started | 0 (Participants did not enter Stage 2 of the study.) | 0 (Participants did not enter Stage 2 of the study.) | 0 (Participants did not enter Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 120 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 39 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 40 (Participants who were randomized to Stage 2 of the study.) | 118 (Participants who were randomized to Stage 2 of the study.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 32 | 36 | 37 | 37 | 35 | 38 | 105 | 32 | 34 | 36 | 36 | 36 | 38 | 105 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 8 | 4 | 3 | 3 | 5 | 2 | 15 | 8 | 5 | 4 | 4 | 4 | 2 | 13 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 1 | 0 | 3 | 3 | 1 | 6 | 5 | 1 | 1 | 3 | 3 | 1 | 6 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 3
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Started | 0 | 0 | 0 | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 0 (Participants did not enter Stage 3 of the study.) | 108 (Participants who were randomized to Stage 3 of the study.) | 108 (Participants who were randomized to Stage 3 of the study.) | 104 (Participants who were randomized to Stage 3 of the study.) | 105 (Participants who were randomized to Stage 3 of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 91 | 88 | 86 | 87
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 20 | 18 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 7 | 4
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received a primary or booster dose of GBS6 vaccine or placebo.
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 microgram of Group B Streptococcus 6-valent (GBS6) vaccine with aluminium phosphate, intramuscularly on Day 1.
- Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 1: Placebo (Nonpregnant): Non pregnant participants were randomized to receive placebo (saline control) intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant) | Total
Number analyzed (Participants) | 22 | 22 | 22 | 40 | 40 | 40 | 40 | 40 | 40 | 120 | 40 | 39 | 40 | 40 | 40 | 40 | 118 | 108 | 108 | 104 | 105 | 1208
Age, Customized [Count of Participants; unit: Participants]
  Full term newborn infants (Gestational age >= 37 weeks) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 36 | 39 | 40 | 39 | 39 | 116 | 0 | 0 | 95 | 98 | 539
  Preterm newborn infants (Gestational age <37 weeks) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 8 | 6 | 25
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  18-40 Years | 22 | 22 | 22 | 40 | 40 | 40 | 40 | 40 | 40 | 120 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 | 108 | 0 | 0 | 642
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 22 | 40 | 40 | 40 | 40 | 40 | 40 | 120 | 17 | 20 | 19 | 20 | 26 | 21 | 55 | 108 | 108 | 60 | 54 | 934
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 19 | 21 | 20 | 14 | 19 | 63 | 0 | 0 | 44 | 51 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 22 | 22 | 22 | 40 | 40 | 40 | 40 | 40 | 40 | 120 | 40 | 39 | 40 | 40 | 40 | 40 | 118 | 82 | 80 | 78 | 78 | 1101
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4
  Race: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 24 | 23 | 22 | 92
  Race: Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 6
  Race: Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic/non-Latino | 22 | 22 | 22 | 40 | 40 | 40 | 40 | 40 | 40 | 120 | 40 | 39 | 40 | 40 | 40 | 40 | 118 | 100 | 102 | 96 | 99 | 1180
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6 | 8 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Primary Dose: Non-Pregnant Participants Stage 1
Description: Local reactions (redness, swelling, and pain at the injection site of the left arm) were recorded by participants in e-diary. Erythema/Redness and induration/swelling were measured and recorded in measuring device units (1 measuring device unit=0.5 centimeter [cm]). Grading: Grade 1/mild (greater than [>] 2.5 to 5.0 cm), Grade 2/moderate (>5.0 to 10.0 cm), Grade 3/severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as Grade 1/mild (did not interfere with activity), Grade2/moderate (interfered with activity), Grade 3/severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7 after Primary Dose
Population: Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a primary of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant)
Number analyzed (Participants) | 22 | 22 | 22
Percentage of Participants
  Pain at injection site (Any) | 27.3 [10.7 to 50.2] | 27.3 [10.7 to 50.2] | 13.6 [2.9 to 34.9]
  Pain at injection site (Mild) | 22.7 [7.8 to 45.4] | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2]
  Pain at injection site (Moderate) | 4.5 [0.1 to 22.8] | 13.6 [2.9 to 34.9] | 4.5 [0.1 to 22.8]
  Pain at injection site (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Pain at injection site (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Erythema/redness (Any) | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8]
  Erythema/redness (Mild) | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8]
  Erythema/redness (Moderate) | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Erythema/redness (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Erythema/redness (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Induration/swelling (Any) | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2] | 0 [0.0 to 15.4]
  Induration/swelling (Mild) | 9.1 [1.1 to 29.2] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Induration/swelling (Moderate) | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Induration/swelling (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Induration/swelling (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]

2. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Booster Dose: Non-Pregnant Women Stage 1
Description: as for outcome 1
Time Frame: Day 1 (day of vaccination) to Day 7 after booster dose
Population: Safety analysis set included all participants who received a booster dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant): Non pregnant participants were randomized to receive a booster dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly at least 2 years after Vaccination 1 on Day 1. Participants were categorized based on their primary dose of GBS6 vaccine with AlPO4.
- Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant): Non pregnant participants were randomized to receive a booster dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly at least 2 years after Vaccination 1 on Day 1. Participants were categorized based on their primary dose of GBS6 vaccine without AlPO4.
- Stage 1 Booster: Placebo (Nonpregnant): Non pregnant participants were randomized to receive a booster dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly at least 2 years after Vaccination 1 on Day 1. Participants were categorized based on their primary dose of Placebo.
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 8
Percentage of Participants
  Pain at injection site (Any) | 72.7 [39.0 to 94.0] | 28.6 [3.7 to 71.0] | 50.0 [15.7 to 84.3]
  Pain at injection site (Mild) | 45.5 [16.7 to 76.6] | 28.6 [3.7 to 71.0] | 37.5 [8.5 to 75.5]
  Pain at injection site (Moderate) | 27.3 [6.0 to 61.0] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]
  Pain at injection site (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Pain at injection site (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Erythema/redness (Any) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Erythema/redness (Mild) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Erythema/redness (Moderate) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Erythema/redness (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Erythema/redness (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Induration/swelling (Any) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Induration/swelling (Mild) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Induration/swelling (Moderate) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Induration/swelling (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Induration/swelling (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]

3. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Primary Dose: Non-Pregnant Participants Stage 1
Description: Systemic events were recorded in e-diary. Fever: oral temperature greater than or equal to (>=) 38.0 degree Celsius (deg C) and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Nausea/vomiting was graded as: Grade 1/mild (1-2 times in 24 hours [h]), Grade 2/moderate: (>2 times in 24h), Grade 3/severe (required intravenous hydration) and Grade 4 (ER visit/hospitalization for hypotensive shock). Diarrhea was graded as: Grade 1/mild (2-3 loose stools in 24h), Grade 2/moderate (4-5 loose stools in 24h), Grade 3/severe (6 or more loose stools in 24h) and Grade 4 (ER visit/hospitalization for severe diarrhea). Fatigue/tiredness, headache, muscle pain and joint pain were graded as: Grade 1/mild (did not interfere with activity), Grade 2/moderate (some interference with activity), Grade 3/severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7 after primary dose
Population: Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant)
Number analyzed (Participants) | 22 | 22 | 22
Percentage of Participants
  Fever (>=38.0 deg C) | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Fever (38.0 to 38.4 deg C) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Fever (38.5 to 38.9 deg C) | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Fever (39.0 to 40.0 deg C) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Fever (>40.0 deg C) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Nausea/vomiting (Any) | 4.5 [0.1 to 22.8] | 9.1 [1.1 to 29.2] | 27.3 [10.7 to 50.2]
  Nausea/vomiting (Mild) | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 9.1 [1.1 to 29.2]
  Nausea/vomiting (Moderate) | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 18.2 [5.2 to 40.3]
  Nausea/vomiting (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Nausea/vomiting (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Diarrhea (Any) | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2] | 18.2 [5.2 to 40.3]
  Diarrhea (Mild) | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2] | 13.6 [2.9 to 34.9]
  Diarrhea (Moderate) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 4.5 [0.1 to 22.8]
  Diarrhea (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Diarrhea (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Headache (Any) | 36.4 [17.2 to 59.3] | 40.9 [20.7 to 63.6] | 50.0 [28.2 to 71.8]
  Headache (Mild) | 31.8 [13.9 to 54.9] | 18.2 [5.2 to 40.3] | 31.8 [13.9 to 54.9]
  Headache (Moderate) | 4.5 [0.1 to 22.8] | 22.7 [7.8 to 45.4] | 13.6 [2.9 to 34.9]
  Headache (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Headache (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Fatigue/tiredness (Any) | 31.8 [13.9 to 54.9] | 31.8 [13.9 to 54.9] | 40.9 [20.7 to 63.6]
  Fatigue/tiredness (Mild) | 18.2 [5.2 to 40.3] | 22.7 [7.8 to 45.4] | 31.8 [13.9 to 54.9]
  Fatigue/tiredness (Moderate) | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2]
  Fatigue/tiredness (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [00 to 15.4]
  Fatigue/tiredness (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Muscle pain (Any) | 4.5 [0.1 to 22.8] | 22.7 [7.8 to 45.4] | 22.7 [7.8 to 45.4]
  Muscle pain (Mild) | 4.5 [0.1 to 22.8] | 13.6 [2.9 to 34.9] | 18.2 [5.2 to 40.3]
  Muscle pain (Moderate) | 0 [0.0 to 15.4] | 9.1 [1.1 to 29.2] | 4.5 [0.1 to 22.8]
  Muscle pain (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Muscle pain (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Joint Pain (Any) | 9.1 [1.1 to 29.2] | 18.2 [5.2 to 40.3] | 4.5 [0.1 to 22.8]
  Joint Pain (Mild) | 9.1 [1.1 to 29.2] | 13.6 [2.9 to 34.9] | 4.5 [0.1 to 22.8]
  Joint Pain (Moderate) | 0 [00 to 15.4] | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4]
  Joint Pain (Severe) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]
  Joint Pain (Grade 4) | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4]

4. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Booster Dose: Non-Pregnant Participants Stage 1
Description: as for outcome 3
Time Frame: Day 1 (day of vaccination) to Day 7 after booster dose
Population: Safety analysis set included all participants who received a booster dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 8
Percentage of Participants
  Fever (38.0 deg C) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fever (38.0 to 38.4 deg C) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fever (38.5 to 38.9 deg C) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fever (39.0 to 40.0 deg C) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fever (>40.0 deg C) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Nausea/vomiting (Any) | 9.1 [0.2 to 41.3] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1]
  Nausea/vomiting (Mild) | 0 [0.0 to 28.5] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1]
  Nausea/vomiting (Moderate) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Nausea/vomiting (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Nausea/vomiting (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Diarrhea (Any) | 18.2 [2.3 to 51.8] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]
  Diarrhea (Mild) | 18.2 [2.3 to 51.8] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Diarrhea (Moderate) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]
  Diarrhea (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Diarrhea (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Headache (Any) | 27.3 [6.0 to 61.0] | 14.3 [0.4 to 57.9] | 62.5 [24.5 to 91.5]
  Headache (Mild) | 0 [0.0 to 28.5] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1]
  Headache (Moderate) | 27.3 [6.0 to 61.0] | 0 [0.0 to 41.0] | 37.5 [8.5 to 75.5]
  Headache (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Headache (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fatigue/tiredness (Any) | 27.3 [6.0 to 61.0] | 0 [0.0 to 41.0] | 37.5 [8.5 to 75.5]
  Fatigue/tiredness (Mild) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fatigue/tiredness (Moderate) | 18.2 [2.3 to 51.8] | 0 [0.0 to 41.0] | 37.5 [8.5 to 75.5]
  Fatigue/tiredness (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Fatigue/tiredness (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Muscle pain (Any) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 37.5 [8.5 to 75.5]
  Muscle pain (Mild) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 25.0 [3.2 to 65.1]
  Muscle pain (Moderate) | 9.1 [0.2 to 41.3] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]
  Muscle pain (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Muscle pain (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Joint Pain (Any) | 18.2 [2.3 to 51.8] | 14.3 [0.4 to 57.9] | 12.5 [0.3 to 52.7]
  Joint Pain (Mild) | 0 [0.0 to 28.5] | 14.3 [0.4 to 57.9] | 0 [0.0 to 36.9]
  Joint Pain (Moderate) | 18.2 [2.3 to 51.8] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]
  Joint Pain (Severe) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]
  Joint Pain (Grade 4) | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]

5. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Through 1 Month After Primary Dose: Non-Pregnant Participants Stage 1
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. Examples of AEs included but were not limited to abnormal test findings; clinically significant signs and symptoms; changes in physical examination findings; hypersensitivity; progression/worsening of underlying disease; drug abuse; drug dependency.
Time Frame: Day 1 (day of vaccination) through 1 Month post primary dose
Population: Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Non pregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant): Non pregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant)
Number analyzed (Participants) | 22 | 22 | 22
Percentage of Participants | 54.5 [32.2 to 75.6] | 45.5 [24.4 to 67.8] | 36.4 [17.2 to 59.3]

6. Primary Outcome: Percentage of Participants Reporting AEs Through 1 Month After Booster Dose: Non-Pregnant Participants Stage 1
Description: as for outcome 5
Time Frame: Day 1 (day of vaccination) through 1 Month post booster dose
Population: Safety analysis set included all participants who received a booster dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 8
Percentage of Participants | 18.2 [2.3 to 51.8] | 0 [0.0 to 41.0] | 12.5 [0.3 to 52.7]

7. Primary Outcome: Percentage of Participants Reporting Medically Attended Adverse Events (MAEs) Through 6 Months After Primary Dose: Non-Pregnant Participants Stage 1
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. Examples of AEs included but were not limited to abnormal test findings; clinically significant signs and symptoms; changes in physical examination findings; hypersensitivity; progression/worsening of underlying disease; drug abuse; drug dependency. A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: Day 1 (day of vaccination) through 6 Months post primary dose
Population: Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant)
Number analyzed (Participants) | 22 | 22 | 22
Percentage of Participants | 45.5 [24.4 to 67.8] | 40.9 [20.7 to 63.6] | 40.9 [20.7 to 63.6]

8. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) Through 6 Months After Primary Dose: Non-Pregnant Participants Stage 1
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. Examples of AEs included but were not limited to abnormal test findings; clinically significant signs and symptoms; changes in physical examination findings; hypersensitivity; progression/worsening of underlying disease; drug abuse; drug dependency. A SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: Day 1 (day of vaccination) through 6 Months post primary dose
Population: Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant); Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant)
Number analyzed (Participants) | 22 | 22 | 22
Percentage of Participants | 0 [0.0 to 15.4] | 0 [00 to 15.4] | 0 [0.0 to 15.4]

9. Primary Outcome: Percentage of Participants Reporting MAEs Approximately 7 to 12 Months After Booster Dose: Non-Pregnant Participants Stage 1
Description: as for outcome 7
Time Frame: Day 1 (day of vaccination) through approximately 7 to 12 months post booster dose
Population: Safety analysis set included all participants who received a booster dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 8
Percentage of Participants | 0 [0.0 to 28.5] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1]

10. Primary Outcome: Percentage of Participants Reporting SAEs Approximately 7 to 12 Months After Booster Dose: Non-Pregnant Participants Stage 1
Description: as for outcome 8
Time Frame: Day 1 (day of vaccination) through approximately 7 to 12 months post booster dose
Population: Safety analysis set included all participants who received a booster dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 8
Percentage of Participants | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]

11. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities at 2 Week Follow-up Visit: Maternal Participants Stage 2
Description: Hemoglobin: Grade 1, Platelets High: Grade 2, White blood cells decreased: Grade 1, Neutrophils (Absolute): Grade 1, Basophils (Absolute): Grade 2, Lymphocytes Low (Absolute): Grade1, Blood urea nitrogen (bun): Grade 1, Aspartate aminotransferase (AST): Grade 2, Alanine aminotransferase (ALT): Grade 1 and 3 and Alkaline phosphate: Grade 1. Grades were considered as 1: mild, 2: moderate, 3: severe. Only categories with non-zero values were reported for this outcome measure.
Time Frame: 2 weeks after vaccination in Stage 2
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo. Here , number of participants analyzed signifies number of participants in the sentinel cohort (subset of Stage 2 maternal participants) evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 14 | 12 | 42
Percentage of Participants
  Hemoglobin Grade 1 | 0 | 7.1 | 0 | 7.1 | 0 | 0 | 2.4
  Platelets High Grade 2 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0
  White blood cells decreased Grade 1 | 15.4 | 21.4 | 7.1 | 0 | 0 | 8.3 | 7.1
  Neutrophils (Absolute) Grade 1 | 7.7 | 35.7 | 7.1 | 21.4 | 7.1 | 0 | 9.5
  Basophils (Absolute) Grade 2 | 0 | 0 | 14.3 | 21.4 | 7.1 | 0 | 2.4
  Lymphocytes Low (Absolute) Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2.4
  Blood urea nitrogen Grade 1 | 1 | 7.1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2.4
  Alanine aminotransferase Grade 1 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2.4
  Alkaline phosphate Grade 1 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0

12. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination: Maternal Participants Stage 2
Description: Local reactions (redness, swelling, and pain at the injection site of the left arm) were recorded by participants in e-diary. Erythema/Redness and induration/swelling were measured and recorded in measuring device units (1 measuring device unit=0.5 cm). Grading: Grade 1/mild (> 2.5 to 5.0 cm), Grade 2/moderate (>5.0 to 10.0 cm), Grade 3/severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as Grade 1/mild (did not interfere with activity), Grade2/moderate (interfered with activity), Grade 3/severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7 after Vaccination
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo. Here, number analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 39 | 40 | 40 | 120
Percentage of Participants
  Pain at injection site (Any) | 37.5 [22.7 to 54.2] | 15.0 [5.7 to 29.8] | 40.0 [24.9 to 56.7] | 15.4 [5.9 to 30.5] | 47.5 [31.5 to 63.9] | 35.0 [20.6 to 51.7] | 15.8 [9.8 to 23.6]
  Pain at injection site (Mild) | 32.5 [18.6 to 49.1] | 12.5 [4.2 to 26.8] | 35.0 [20.6 to 51.7] | 15.4 [5.9 to 30.5] | 42.5 [27.0 to 59.1] | 20.0 [9.1 to 35.6] | 12.5 [7.2 to 19.8]
  Pain at injection site (Moderate) | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 0 [0.0 to 9.0] | 5.0 [0.6 to 16.9] | 15.0 [5.7 to 29.8] | 3.3 [0.9 to 8.3]
  Pain at injection site (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Pain at injection site (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Erythema/redness (Any) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.5 [0.01 to 13.2] | 0 [0.0 to 9.0] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 1.7 [0.2 to 5.9]
  Erythema/redness (Mild) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 0.8 [0.0 to 4.6]
  Erythema/redness (Moderate) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Erythema/redness (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Erythema/redness (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Induration/swelling (Any) | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 2.6 [0.1 to 13.5] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 0.8 [0.0 to 4.6]
  Induration/swelling (Mild) | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 0 [0.0 to 3.0]
  Induration/swelling (Moderate) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Induration/swelling (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Induration/swelling (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]

13. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination: Maternal Participants Stage 3
Description: as for outcome 12
Time Frame: Day 1 (day of vaccination) to Day 7 after Vaccination
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Stage 3: GBS6 20 mcg Without AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 106 | 103
Percentage of Participants
  Pain at injection site (Any) | 30.2 [21.7 to 39.9] | 18.4 [11.5 to 27.3]
  Pain at injection site (Mild) | 25.5 [17.5 to 34.9] | 13.6 [7.6 to 21.8]
  Pain at injection site (Moderate) | 4.7 [1.5 to 10.7] | 4.9 [1.6 to 11.0]
  Pain at injection site (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Pain at injection site (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Erythema/redness (Any) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Erythema/redness (Mild) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Erythema/redness (Moderate) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Erythema/redness (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Erythema/redness (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Induration/swelling (Any) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Induration/swelling (Mild) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Induration/swelling (Moderate) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Induration/swelling (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Induration/swelling (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]

14. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days Following Administration of Investigational Product: Maternal Participants Stage 2
Description: Systemic events were recorded in e-diary. Fever: oral temperature >=38.0 deg C and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Nausea/vomiting was graded as: Grade 1/mild (1-2 times in 24 h), Grade 2/moderate: (>2 times in 24h), Grade 3/severe (required intravenous hydration) and Grade 4 (ER visit/hospitalization for hypotensive shock). Diarrhea was graded as: Grade 1/mild (2-3 loose stools in 24h), Grade 2/moderate (4-5 loose stools in 24h), Grade 3/severe (6 or more loose stools in 24h) and Grade 4 (ER visit/hospitalization for severe diarrhea). Fatigue/tiredness, headache, muscle pain and joint pain were graded as: Grade 1/mild (did not interfere with activity), Grade 2/moderate (some interference with activity), Grade 3/severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7 after Vaccination
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 39 | 40 | 40 | 120
Percentage of Participants
  Fever (>=38.0 deg C) | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 7.7 [1.6 to 20.9] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 5.0 [1.9 to 10.6]
  Fever (38.0 to 38.4 deg C) | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 5.1 [0.6 to 17.3] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 3.3 [0.9 to 8.3]
  Fever (38.5 to 38.9 deg C) | 0 [0.0 to 8.8] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 1.7 [0.2 to 5.9]
  Fever (39.0 to 40.0 deg C) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Fever (>40.0 deg C) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Nausea/vomiting (Any) | 15.0 [5.7 to 29.8] | 7.5 [1.6 to 20.4] | 20.0 [9.1 to 35.6] | 15.4 [5.9 to 30.5] | 15.0 [5.7 to 29.8] | 22.5 [10.8 to 38.5] | 26.7 [19.0 to 35.5]
  Nausea/vomiting (Mild) | 10.0 [2.8 to 23.7] | 5.0 [0.6 to 16.9] | 17.5 [7.3 to 32.8] | 10.3 [2.9 to 242] | 12.5 [4.2 to 26.8] | 17.5 [7.3 to 32.8] | 19.2 [12.6 to 27.4]
  Nausea/vomiting (Moderate) | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 5.1 [0.6 to 17.3] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 7.5 [3.5 to 13.8]
  Nausea/vomiting (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Nausea/vomiting (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [00 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Diarrhea (Any) | 5.0 [0.6 to 16.9] | 17.5 [7.3 to 32.8] | 10.0 [2.8 to 23.7] | 23.1 [11.1 to 39.3] | 7.5 [1.6 to 20.4] | 10.0 [2.8 to 23.7] | 16.7 [10.5 to 24.6]
  Diarrhea (Mild) | 5.0 [0.6 to 16.9] | 12.5 [4.2 to 26.8] | 7.5 [1.6 to 20.4] | 7.7 [1.6 to 20.9] | 7.5 [1.6 to 20.4] | 10.0 [2.8 to 23.7] | 15.0 [9.1 to 22.7]
  Diarrhea (Moderate) | 0 [0.0 to 8.8] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 12.8 [4.3 to 27.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Diarrhea (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Diarrhea (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Headache (Any) | 30.0 [16.6 to 46.5] | 47.5 [31.5 to 63.9] | 30.0 [16.6 to 46.5] | 33.3 [19.1 to 50.2] | 32.5 [18.6 to 49.1] | 40.0 [24.9 to 56.7] | 33.3 [25.0 to 42.5]
  Headache (Mild) | 22.5 [10.8 to 38.5] | 37.5 [22.7 to 54.2] | 15.0 [5.7 to 29.8] | 17.9 [7.5 to 33.5] | 25.0 [12.7 to 41.2] | 22.5 [10.8 to 38.5] | 25.0 [17.5 to 33.7]
  Headache (Moderate) | 7.5 [1.6 to 20.4] | 10.0 [2.8 to 23.7] | 15.0 [5.7 to 29.8] | 15.4 [5.9 to 30.5] | 7.5 [1.6 to 20.4] | 17.5 [7.3 to 32.8] | 7.5 [3.5 to 13.8]
  Headache (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Headache (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Fatigue/tiredness (Any) | 37.5 [22.7 to 54.2] | 45.0 [29.3 to 61.5] | 37.5 [22.7 to 54.2] | 38.5 [23.4 to 55.4] | 47.5 [31.5 to 63.9] | 42.5 [27.0 to 59.1] | 40.0 [31.2 to 49.3]
  Fatigue/tiredness (Mild) | 27.5 [14.6 to 43.9] | 22.5 [10.8 to 38.5] | 25.0 [12.7 to 41.2] | 17.9 [7.5 to 33.5] | 35.0 [20.6 to 51.7] | 30.0 [16.6 to 46.5] | 23.3 [16.1 to 31.9]
  Fatigue/tiredness (Moderate) | 10.0 [2.8 to 23.7] | 22.5 [10.8 to 38.5] | 12.5 [4.2 to 26.8] | 17.9 [7.5 to 33.5] | 10.0 [2.8 to 23.7] | 12.5 [4.2 to 26.8] | 14.2 [8.5 to 21.7]
  Fatigue/tiredness (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 2.5 [0.5 to 7.1]
  Fatigue/tiredness (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Muscle pain (Any) | 12.5 [4.2 to 26.8] | 25.0 [12.7 to 41.2] | 17.5 [7.3 to 32.8] | 15.4 [5.9 to 30.5] | 17.5 [7.3 to 32.8] | 25.0 [12.7 to 41.2] | 15.8 [9.8 to 23.6]
  Muscle pain (Mild) | 7.5 [1.6 to 20.4] | 12.5 [4.2 to 26.8] | 15.0 [5.7 to 29.8] | 10.3 [2.9 to 24.2] | 12.5 [4.2 to 26.8] | 12.5 [4.2 to 26.8] | 10.8 [5.9 to 17.8]
  Muscle pain (Moderate) | 5.0 [0.6 to 16.9] | 12.5 [4.2 to 26.8] | 2.5 [0.1 to 13.2] | 5.1 [0.6 to 17.3] | 2.5 [0.1 to 13.2] | 12.5 [4.2 to 26.8] | 5.0 [1.9 to 10.6]
  Muscle pain (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Muscle pain (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Joint pain (Any) | 10.0 [2.8 to 23.7] | 10.0 [2.8 to 23.7] | 2.5 [0.1 to 13.2] | 12.8 [4.3 to 27.4] | 15.0 [5.7 to 29.8] | 20.0 [9.1 to 35.6] | 16.7 [10.5 to 24.6]
  Joint pain (Mild) | 7.5 [1.6 to 20.4] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 7.7 [1.6 to 20.9] | 10.0 [2.8 to 23.7] | 10.0 [2.8 to 23.7] | 11.7 [6.5 to 18.8]
  Joint pain (Moderate) | 2.5 [0.1 to 13.2] | 7.5 [1.6 to 20.4] | 0 [0.0 to 8.8] | 5.1 [0.6 to 17.3] | 2.5 [0.1 to 13.2] | 10.0 [2.8 to 23.7] | 5.0 [1.9 to 10.6]
  Joint pain (Severe) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]
  Joint pain (Grade 4) | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.0]

15. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days Following Administration of Investigational Product: Maternal Participants Stage 3
Description: as for outcome 14
Time Frame: Day 1 (day of vaccination) to Day 7 after Vaccination
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 106 | 103
Percentage of Participants
  Fever (>=38.0 deg C) | 2.8 [0.6 to 8.0] | 4.9 [1.6 to 11.0]
  Fever (38.0 to 38.4 deg C) | 2.8 [0.6 to 8.0] | 2.9 [0.6 to 8.3]
  Fever (38.5 to 38.9 deg C) | 0 [0.0 to 3.4] | 1.9 [0.2 to 6.8]
  Fever (39.0 to 40.0 deg C) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Fever (>40.0 deg C) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Nausea/vomiting (Any) | 21.7 [14.3 to 30.8] | 29.1 [20.6 to 38.9]
  Nausea/vomiting (Mild) | 18.9 [11.9 to 27.6] | 22.3 [14.7 to 31.6]
  Nausea/vomiting (Moderate) | 2.8 [0.6 to 8.0] | 6.8 [2.8 to 13.5]
  Nausea/vomiting (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Nausea/vomiting (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Diarrhea (Any) | 12.3 [6.7 to 20.1] | 11.7 [6.2 to 19.5]
  Diarrhea (Mild) | 12.3 [6.7 to 20.1] | 8.7 [4.1 to 15.9]
  Diarrhea (Moderate) | 0 [0.0 to 3.4] | 2.9 [0.6 to 8.3]
  Diarrhea (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Diarrhea (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Headache (Any) | 36.8 [27.6 to 46.7] | 37.9 [28.5 to 48.0]
  Headache (Mild) | 19.8 [12.7 to 28.7] | 30.1 [21.5 to 39.9]
  Headache (Moderate) | 17.0 [10.4 to 25.5] | 7.8 [3.4 to 14.7]
  Headache (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Headache (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Fatigue/tiredness (Any) | 42.5 [32.9 to 52.4] | 42.7 [33.0 to 52.8]
  Fatigue/tiredness (Mild) | 24.5 [16.7 to 33.8] | 24.3 [16.4 to 33.7]
  Fatigue/tiredness (Moderate) | 17.9 [11.2 to 26.6] | 15.5 [9.1 to 24.0]
  Fatigue/tiredness (Severe) | 0 [0.0 to 3.4] | 2.9 [0.6 to 8.3]
  Fatigue/tiredness (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Muscle pain (Any) | 18.9 [11.9 to 27.6] | 14.6 [8.4 to 22.9]
  Muscle pain (Mild) | 13.2 [7.4 to 21.2] | 5.8 [2.2 to 12.2]
  Muscle pain (Moderate) | 5.7 [2.1 to 11.9] | 8.7 [4.1 to 15.9]
  Muscle pain (Severe) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Muscle pain (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]
  Joint pain (Any) | 15.1 [8.9 to 23.4] | 13.6 [7.6 to 21.8]
  Joint pain (Mild) | 9.4 [4.6 to 16.7] | 8.7 [4.1 to 15.9]
  Joint pain (Moderate) | 5.7 [2.1 to 11.9] | 3.9 [1.1 to 9.6]
  Joint pain (Severe) | 0 [0.0 to 3.4] | 1.0 [0.0 to 5.3]
  Joint pain (Grade 4) | 0 [0.0 to 3.4] | 0 [0.0 to 3.5]

16. Primary Outcome: Percentage of Participants Reporting AEs Through 1 Month After Administration of Investigational Product: Maternal Participants Stage 2
Description: as for outcome 5
Time Frame: Day 1 (day of vaccination) through 1 Month post vaccination
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 120
Percentage of Participants | 27.5 [14.6 to 43.9] | 40.0 [24.9 to 56.7] | 22.5 [10.8 to 38.5] | 22.5 [10.8 to 38.5] | 30.0 [16.6 to 46.5] | 30.0 [16.6 to 46.7] | 27.5 [19.7 to 36.7]

17. Primary Outcome: Percentage of Participants Reporting AEs Through 1 Month After Administration of Investigational Product: Maternal Participants Stage 3
Description: as for outcome 5
Time Frame: Day 1 (day of vaccination) through 1 Month post vaccination
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 108 | 108
Percentage of Participants | 36.1 [27.1 to 45.9] | 32.4 [23.7 to 42.1]

18. Primary Outcome: Percentage of Participants With SAEs From Day 1 Through 12 Months Post-delivery: Maternal Participants Stage 2
Description: as for outcome 8
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 120
Percentage of Participants | 17.5 [7.3 to 32.8] | 45.0 [29.3 to 61.5] | 22.5 [0.8 to 38.5] | 27.5 [14.6 to 43.9] | 20.0 [9.1 to 35.6] | 35.0 [20.6 to 51.7] | 25.0 [17.5 to 33.7]

19. Primary Outcome: Percentage of Participants With SAEs From Day 1 Through 12 Months Post-delivery: Maternal Participants Stage 3
Description: as for outcome 8
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 108 | 108
Percentage of Participants | 19.4 [12.5 to 28.2] | 21.3 [14.0 to 30.2]

20. Primary Outcome: Percentage of Participants With MAEs From Day 1 Through 12 Months Post-delivery: Maternal Participants Stage 2
Description: as for outcome 7
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 120
Percentage of Participants | 30.0 [16.6 to 46.5] | 45.0 [29.3 to 61.5] | 30.0 [16.6 to 46.5] | 27.5 [14.6 to 43.9] | 25.0 [12.7 to 41.2] | 32.5 [18.6 to 49.1] | 42.5 [33.5 to 51.9]

21. Primary Outcome: Percentage of Participants With MAEs From Day 1 Through 12 Months Post-delivery: Maternal Participants Stage 3
Description: as for outcome 7
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 108 | 108
Percentage of Participants | 51.9 [42.0 to 61.6] | 42.6 [33.1 to 52.5]

22. Primary Outcome: Percentage of Participants With Obstetric Complications From Visit 1 Through 12 Months Post-delivery: Maternal Participants Stage 2
Description: Obstetric complications such as: prepartum period, intrapartum period and postpartum period were reported in this outcome measure.
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 120
Percentage of Participants
  Prepartum Period | 5.0 [0.6 to 16.9] | 12.5 [4.2 to 26.8] | 5.0 [0.6 to 16.9] | 10.0 [2.8 to 23.7] | 5.0 [0.6 to 16.9] | 10.0 [2.8 to 23.7] | 11.7 [6.5 to 18.8]
  Intrapartum Period | 10.0 [2.8 to 23.7] | 30.0 [16.6 to 46.5] | 10.0 [2.8 to 23.7] | 15.0 [5.7 to 29.8] | 10.0 [2.8 to 23.7] | 20.0 [9.1 to 35.6] | 11.7 [6.5 to 18.8]
  Postpartum Period | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 1.7 [0.2 to 5.9]

23. Primary Outcome: Percentage of Participants With Obstetric Complications From Day 1 Through 12 Months Post-delivery: Maternal Participants Stage 3
Description: as for outcome 22
Time Frame: Day 1 (day of vaccination) through 12 Month post delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 108 | 108
Percentage of Participants
  Prepartum Period | 9.3 [4.5 to 16.4] | 13.0 [7.3 to 20.8]
  Intrapartum Period | 13.9 [8.0 to 21.9] | 13.0 [7.3 to 20.8]
  Postpartum Period | 2.8 [0.6 to 7.9] | 1.9 [0.2 to 6.5]

24. Primary Outcome: Percentage of Participants With Each Delivery Outcome and Delivery Mode: Maternal Participants Stage 2
Description: Delivery Outcome included full term live delivery, premature live delivery, Stillbirth, induced/elective abortion and unknown. Mode of delivery included: vaginal delivery, Cesarean section: elective, semi-elective and emergency were reported in this outcome measure.
Time Frame: At delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 120
Percentage of Participants
  Full term live delivery | 92.5 | 90.0 | 97.5 | 100.0 | 97.5 | 97.5 | 95.8
  Premature live delivery | 7.5 | 7.5 | 2.5 | 0 | 2.5 | 2.5 | 2.5
  Stillbirth | 0 | 2.5 | 0 | 0 | 0 | 0 | 0
  Induced/elective abortion | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Delivery outcome-Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1.7
  Vaginal delivery | 85.0 | 60.0 | 82.5 | 67.5 | 82.5 | 70.0 | 76.7
  Cesarean section: elective | 5.0 | 12.5 | 7.5 | 5.0 | 5.0 | 10.0 | 8.3
  Cesarean section: semi-elective | 0 | 0 | 0 | 0 | 0 | 0 | 0.8
  Cesarean section: emergency | 10.0 | 27.5 | 10.0 | 27.5 | 12.5 | 20.0 | 12.5
  Delivery mode-Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1.7

25. Primary Outcome: Percentage of Participants With Each Delivery Outcome and Delivery Mode: Maternal Participants Stage 3
Description: as for outcome 24
Time Frame: At delivery
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 108 | 108
Percentage of Participants
  Full term live delivery | 88.0 | 91.7
  Premature live delivery | 7.4 | 5.6
  Stillbirth | 0.9 | 0
  Induced/elective abortion | 0 | 0
  Delivery outcome-Unknown | 3.7 | 2.7
  Vaginal delivery | 72.2 | 75.9
  Cesarean section: elective | 12.0 | 9.3
  Cesarean section: semi-elective | 1.9 | 0
  Cesarean section: emergency | 10.2 | 12.0
  Delivery mode-Unknown | 3.7 | 2.8

26. Primary Outcome: Percentage of Participants With Gestational Age at Birth: Infant Participants Stage 2
Description: Gestational age of participants at birth in weeks included: greater than or equal to (>=)24 weeks to less than (<) 28 weeks, >=28 weeks to <34 weeks, >=34 weeks to <37 weeks, >=37 weeks to <42 weeks, >=42 weeks.
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Percentage of Participants
  >=24 weeks to <28 weeks | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=28 weeks to <34 weeks | 2.5 | 2.6 | 0 | 0 | 0 | 0 | 0
  >=34 weeks to <37 weeks | 5.0 | 5.1 | 2.5 | 0 | 2.5 | 2.5 | 1.7
  >=37 weeks to <42 weeks | 87.5 | 84.6 | 97.5 | 92.5 | 95.0 | 95.0 | 94.9
  >=42 weeks | 5.0 | 7.7 | 0 | 7.5 | 2.5 | 2.5 | 3.4

27. Primary Outcome: Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score at 1 Minute: Infant Participants Stage 2
Description: APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low. APGAR score at 1 minute were reported in this outcome measure.
Time Frame: At 1 minute of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Unit on a scale
Groups:
- Stage 2: GBS6 5 mcg With AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 5 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 5 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 5 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg With AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 10 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 10 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 10 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg With AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 2: GBS6 20 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 38 | 40 | 40 | 40 | 40 | 113
Unit on a scale | 9.0 [8 to 9] | 9.0 [6 to 9] | 9.0 [8 to 9] | 9.0 [7 to 9] | 9.0 [3 to 9] | 9.0 [5 to 9] | 9.0 [1 to 9]

28. Primary Outcome: Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score at 5 Minutes: Infant Participants Stage 2
Description: APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low. APGAR score at 5 minute were reported in this outcome measure.
Time Frame: At 5 minutes of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Unit on a scale | 10.0 [8 to 10] | 10.0 [8 to 10] | 10.0 [9 to 10] | 10.0 [9 to 10] | 10.0 [7 to 10] | 10.0 [5 to 10] | 10.0 [4 to 10]

29. Primary Outcome: Number of Participants According to Age Determined by Ballard Score: Infant Participants Stage 2
Description: The Ballard score is a commonly used technique of gestational age assessment. It assists healthcare providers in determining if an infant is premature, on time, or post-term based on physical traits. This scoring allows for the estimation of age in the range of 26 weeks to 44 weeks Participants according to age determined by Ballard score: at <37 weeks 0 days, >=37 weeks to <42 weeks, >=42 weeks were reported in this outcome measure. Ballard score was not conducted routinely/mandatory.
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants
  <37 weeks 0 days | 1 [8 to 10] | 2 [8 to 10] | 1 [9 to 10] | 1 [9 to 10] | 2 [7 to 10] | 2 [5 to 10] | 4 [4 to 10]
  >=37 weeks to <42 weeks | 6 | 3 | 7 | 4 | 3 | 4 | 18
  >=42 weeks | 1 | 1 | 1 | 1 | 4 | 0 | 2
  Not reported | 32 | 33 | 31 | 34 | 31 | 34 | 94

30. Primary Outcome: Number of Participants With Newborn Assessment at Birth: Infant Participants Stage 2
Description: Participants with newborn assessment at birth included: normal, congenital malformation/anomaly, other neonatal problem were reported in this outcome measure.
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants
  Normal | 34 [8 to 10] | 30 [8 to 10] | 38 [9 to 10] | 38 [9 to 10] | 34 [7 to 10] | 35 [5 to 10] | 89 [4 to 10]
  Congenital malformation/anomaly | 7 | 8 | 2 | 2 | 5 | 6 | 26
  Other neonatal problem | 3 | 4 | 2 | 2 | 2 | 4 | 5

31. Primary Outcome: Number of Participants With Vital Status: Infant Participants Stage 2
Description: Participants according to vital status as: live or neonatal death were reported in this outcome measure.
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants
  Live | 40 [8 to 10] | 38 [8 to 10] | 40 [9 to 10] | 40 [9 to 10] | 40 [7 to 10] | 40 [5 to 10] | 117 [4 to 10]
  Neonatal death | 0 | 1 | 0 | 0 | 0 | 0 | 1

32. Primary Outcome: Number of Participants With Gestational Age of Participants at Birth: Infant Participants Stage 3
Description: as for outcome 26
Time Frame: At 1 minute of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 3: Placebo (Infant): Infant participants born to the maternal participants randomized to receive placebo (saline control) intramuscularly on Day 1.
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants
  >=24 weeks to <28 weeks | 0 | 0
  >=28 weeks to <34 weeks | 1 | 2
  >=34 weeks to <37 weeks | 7 | 4
  >=37 weeks to <42 weeks | 94 | 94
  >=42 weeks | 1 | 4
  Unknown | 1 | 1

33. Primary Outcome: Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score at 1 Minute: Infant Participants Stage 3
Description: APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low. Appearance, pulse, grimace, activity, and respiration (APGAR) score at 1 minute were reported in this outcome measure.
Time Frame: At 1 minute of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Unit on a scale | 9.0 [2 to 10] | 9.0 [1 to 9]

34. Primary Outcome: APGAR Score at 5 Minutes: Infant Participants Stage 3
Description: APGAR is a scoring system that evaluates Activity, Pulse, Grimace, Appearance, and Respiration. Each category is given a score of 0-2 points (with 0 being absent and 2 being normal), the points are then combined for a total score that ranges from 0-10. Scores 7 and above are generally normal, 4 to 6 are fairly low, and 2 and below are considered critically low. Appearance, pulse, grimace, activity, and respiration (APGAR) score at 5 minute were reported in this outcome measure.
Time Frame: At 5 minutes of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Unit on a scale | 10.0 [7 to 10] | 10.0 [4 to 10]

35. Primary Outcome: Number of Participants According to Age Determined by Ballard Score: Infant Participants Stage 3
Description: as for outcome 29
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants
  <37 weeks 0 days | 4 | 4
  >=37 weeks to <42 weeks | 30 | 37
  >=42 weeks | 5 | 4
  Not reported | 65 | 60

36. Primary Outcome: Number of Participants With Newborn Assessment at Birth: Infant Participants Stage 3
Description: as for outcome 30
Time Frame: At 5 minutes of Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants
  Normal | 82 | 79
  Congenital malformation/anomaly | 15 | 16
  Other neonatal problem | 12 | 15

37. Primary Outcome: Number of Participants With Vital Status: Infant Participants Stage 3
Description: Participants according to vital status as: live or neonatal death were reported in this outcome measure.
Time Frame: At Birth
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants
  Live | 103 | 104
  Neonatal death | 1 | 1

38. Primary Outcome: Number of Participants With AEs From Birth to 6 Weeks of Age: Infant Participants Stage 2
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage.
Time Frame: From Birth to 6 Weeks
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants | 26 [8 to 10] | 21 [8 to 10] | 25 [9 to 10] | 21 [9 to 10] | 19 [7 to 10] | 18 [5 to 10] | 68 [4 to 10]

39. Primary Outcome: Numberof Participants With AEs From Birth to 6 Weeks of Age: Infant Participants Stage 3
Description: as for outcome 38
Time Frame: From Birth to 6 Weeks
Population: Safety analysis set included all participants whose mother received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants | 65 | 64

40. Primary Outcome: Number of Participants With SAEs From Birth to 12 Months of Age: Infant Participants Stage 2
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. A SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants whose mothers received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants | 17 [8 to 10] | 19 [8 to 10] | 15 [9 to 10] | 12 [9 to 10] | 19 [7 to 10] | 14 [5 to 10] | 60 [4 to 10]

41. Primary Outcome: Number of Participants With SAEs From Birth to 12 Months of Age: Infant Participants Stage 3
Description: as for outcome 40
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants whose mothers received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants | 45 | 46

42. Primary Outcome: Number of Participants With MAEs From Birth to 12 Months of Age: Infant Participants Stage 2
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility.
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants whose mothers received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants | 22 [8 to 10] | 14 [8 to 10] | 19 [9 to 10] | 21 [9 to 10] | 18 [7 to 10] | 18 [5 to 10] | 58 [4 to 10]

43. Primary Outcome: Number of Participants With MAEs From Birth to 12 Months of Age: Infant Participants Stage 3
Description: as for outcome 42
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Participants | 65 | 66

44. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest From Birth to 12 Months of Age: Infant Participants Stage 2
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention or medical device; the event need not necessarily had a causal relationship with the treatment or usage. AEs of special interest included: major congenital anomalies, developmental delay and suspected or confirmed GBS infection.
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Participants of Participants
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 40 | 39 | 40 | 40 | 40 | 40 | 118
Participants of Participants
  Major congenital anomalies | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 1.7 [0.2 to 6.0]
  Developmental delay | 0 [0.0 to 8.8] | 2.6 [0.1 to 13.5] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0.8 [0.0 to 4.6]
  Suspected or confirmed GBS infection | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 3.1]

45. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest From Birth to 12 Months of Age: Infant Participants Stage 3
Description: as for outcome 44
Time Frame: From Birth to 12 Months
Population: Safety analysis set included all participants who received a dose of GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 104 | 105
Percentage of Participants
  Major congenital anomalies | 0 [0.0 to 3.5] | 0 [0.0 to 3.5]
  Developmental delay | 1.0 [0.0 to 5.2] | 0 [0.0 to 3.5]
  Suspected or confirmed GBS infection | 0 [0.0 to 3.5] | 0 [0.0 to 3.5]

46. Secondary Outcome: Geometric Mean Concentration (GMCs) of Group B Streptococcus (GBS) Serotype-Specific Immunoglobulin G (IgG) at 1 Month After Primary Dose: Non-Pregnant Women Stage 1
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At 1 Month After primary Dose
Population: Evaluable immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Groups:
- Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a primary dose of 20 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
- Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant): Nonpregnant participants were randomized to receive a primary dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
- Stage 1: Placebo (Non Pregnant): Infant participants were randomized to receive placebo (saline control) intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Non Pregnant)
Number analyzed (Participants) | 22 | 22 | 22
microgram per milliliter
  Ia | 64.729 [19.893 to 210.612] | 25.781 [8.040 to 82.661] | 0.152 [0.029 to 0.807]
  Ib | 4.986 [1.639 to 15.165] | 5.546 [1.497 to 20.549] | 0.019 [0.009 to 0.039]
  II | 23.359 [10.941 to 49.870] | 37.920 [14.374 to 100.033] | 0.179 [0.087 to 0.365]
  III | 22.622 [8.569 to 59.725] | 19.065 [8.430 to 43.116] | 0.068 [0.022 to 0.213]
  IV | 5.748 [2.784 to 11.864] | 2.564 [1.292 to 5.091] | 0.041 [0.016 to 0.104]
  V | 0.599 [0.220 to 1.631] | 0.420 [0.105 to 1.676] | 0.058 [0.020 to 0.168]

47. Secondary Outcome: GMCs of GBS Serotype-specific IgG Before and 1 Month, 3 Months, and 6 Months After a Booster Dose: Non Pregnant Women Stage 1
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: Before (immediately before booster vaccination) and at 1, 3 and 6 Months After vaccination as Booster Dose
Population: Evaluable immunogenicity population. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant)
Number analyzed (Participants) | 11 | 7 | 7
microgram per milliliter
  Ia (Before) | 21.088 [5.663 to 78.520] | 3.230 [0.164 to 63.426] | 0.812 [0.026 to 25.244]
  Ia (Month 1) | 86.661 [47.789 to 157.153] | 48.241 [15.580 to 149.375] | 68.222 [3.526 to 1319.87]
  Ia (Month 3) | 60.200 [28.513 to 127.102] | 27.000 [6.370 to 114.442] | 49.958 [3.463 to 720.799]
  Ia (Month 6) | 51.631 [21.557 to 123.660] | 18.936 [4.154 to 86.321] | 23.140 [2.552 to 209.826]
  Ib (Before) | 1.643 [0.457 to 5.914] | 0.215 [0.012 to 3.749] | 0.057 [0.014 to 0.222]
  Ib (Month 1) | 29.416 [17.765 to 48.706] | 11.171 [2.526 to 49.402] | 6.176 [0.928 to 41.110]
  Ib (Month 3) | 16.062 [8.198 to 31.470] | 6.134 [1.183 to 31.813] | 3.479 [0.666 to 18.173]
  Ib (Month 6) | 11.053 [4.697 to 26.010] | 4.033 [0.753 to 21.588] | 2.304 [0.446 to 11.896]
  II (Before) | 4.041 [1.542 to 10.593] | 10.338 [1.123 to 95.149] | 0.185 [0.053 to 0.646]
  II (Month 1) | 113.187 [57.027 to 224.653] | 92.478 [17.542 to 487.530] | 48.523 [10.696 to 220.122]
  II (Month 3) | 64.110 [31.261 to 131.479] | 62.160 [9.893 to 390.578] | 32.569 [6.968 to 152.225]
  II (Month 6) | 38.482 [17.354 to 85.334] | 48.827 [7.872 to 302.837] | 24.262 [5.239 to 112.349]
  III (Before) | 6.765 [1.919 to 23.847] | 3.058 [0.343 to 27.231] | 0.084 [0.017 to 0.403]
  III (Month 1) | 36.579 [17.516 to 76.390] | 30.831 [11.300 to 84.117] | 14.092 [4.614 to 43.045]
  III (Month 3) | 25.006 [11.011 to 56.790] | 18.206 [4.216 to 78.614] | 7.729 [2.486 to 24.024]
  III (Month 6) | 21.808 [9.021 to 52.717] | 12.540 [2.433 to 64.642] | 4.941 [2.015 to 12.117]
  IV (Before) | 0.949 [0.388 to 2.324] | 0.351 [0.080 to 1.545] | 0.031 [0.006 to 0.151]
  IV (Month 1) | 33.784 [18.478 to 61.771] | 14.228 [5.724 to 35.368] | 14.942 [5.920 to 37.717]
  IV (Month 3) | 14.744 [7.275 to 29.882] | 5.820 [2.005 to 16.893] | 7.524 [2.629 to 21.536]
  IV (Month 6) | 9.750 [4.014 to 23.681] | 3.325 [1.082 to 10.218] | 4.918 [1.606 to 15.057]
  V (Before) | 0.245 [0.056 to 1.076] | 0.261 [0.026 to 2.596] | 0.080 [0.012 to 0.532]
  V (Month 1) | 8.208 [2.328 to 28.936] | 7.177 [0.841 to 61.232] | 6.511 [0.665 to 63.696]
  V (Month 3) | 4.454 [1.177 to 16.857] | 3.782 [0.448 to 31.946] | 5.400 [0.710 to 41.094]
  V (Month 6) | 3.086 [0.767 to 12.417] | 2.594 [0.314 to 21.411] | 4.666 [0.601 to 36.239]

48. Secondary Outcome: GMCs of GBS Serotype-specific IgG at 2 Weeks, 1 Month After Vaccination and at Delivery: Maternal Participants Stage 2
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At 2 Weeks after Vaccination, 1 Month After Vaccination and at Delivery
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: microgram per milliliter
Groups:
- Stage 2: GBS6 5 mcg With AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 5 mcg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 39 | 39 | 28 | 26 | 39 | 40 | 103
microgram per milliliter
  Ia (Week 2) | 8.399 [3.031 to 23.274] | 16.089 [7.267 to 35.623] | 11.073 [3.974 to 30.852] | 10.782 [2.432 to 47.800] | 13.813 [4.502 to 42.381] | 41.201 [20.997 to 80.843] | 0.099 [0.055 to 0.178]
  Ia (Month 1) | 8.850 [3.119 to 25.116] | 14.987 [6.881 to 32.640] | 14.356 [4.650 to 44.324] | 16.283 [5.352 to 49.540] | 17.399 [6.456 to 46.894] | 47.200 [29.211 to 76.266] | 0.092 [0.052 to 0.161]
  Ia (At Delivery) | 11.940 [5.566 to 25.613] | 13.901 [5.547 to 34.833] | 14.492 [5.244 to 40.045] | 20.078 [7.642 to 52.750] | 21.991 [8.812 to 54.883] | 39.831 [23.254 to 68.225] | 0.116 [0.063 to 0.211]
  Ib (Week 2) | 0.270 [0.090 to 0.811] | 0.306 [0.106 to 0.878] | 0.315 [0.077 to 1.282] | 1.354 [0.366 to 5.014] | 0.698 [0.315 to 1.548] | 1.245 [0.454 to 3.414] | 0.009 [0.006 to 0.014]
  Ib (Month 1) | 0.275 [0.082 to 0.922] | 0.382 [0.131 to 1.119] | 0.350 [0.098 to 1.248] | 1.102 [0.329 to 3.693] | 0.566 [0.249 to 1.283] | 1.284 [0.491 to 3.362] | 0.009 [0.006 to 0.013]
  Ib (At Delivery) | 0.453 [0.155 to 1.329] | 0.293 [0.101 to 0.847] | 0.625 [0.179 to 2.181] | 1.668 [0.558 to 4.989] | 0.844 [0.388 to 1.838] | 1.388 [0.603 to 3.196] | 0.012 [0.008 to 0.017]
  II (Week 2) | 8.153 [4.325 to 15.368] | 5.294 [2.942 to 9.525] | 8.232 [3.838 to 17.654] | 7.933 [3.596 to 17.498] | 16.009 [7.878 to 32.536] | 22.272 [10.782 to 46.006] | 0.095 [0.067 to 0.135]
  II (Month 1) | 7.784 [3.533 to 17.153] | 4.555 [2.277 to 9.112] | 10.449 [4.742 to 23.026] | 9.691 [5.410 to 17.361] | 12.468 [5.531 to 28.110] | 27.493 [15.334 to 49.295] | 0.112 [0.076 to 0.165]
  II (At Delivery) | 8.676 [4.463 to 16.866] | 3.220 [1.509 to 6.872] | 9.676 [4.528 to 20.679] | 7.158 [3.709 to 13.816] | 15.543 [7.816 to 30.907] | 25.853 [14.640 to 45.655] | 0.139 [0.097 to 0.200]
  III (Week 2) | 1.518 [0.534 to 4.312] | 2.165 [0.829 to 5.658] | 4.164 [1.236 to 14.033] | 2.344 [0.700 to 7.844] | 2.117 [0.847 to 5.296] | 4.979 [1.870 to 13.260] | 0.020 [0.013 to 0.031]
  III (Month 1) | 1.294 [0.432 to 3.878] | 1.638 [0.658 to 4.077] | 7.260 [2.394 to 22.014] | 3.944 [1.428 to 10.895] | 1.627 [0.630 to 4.199] | 5.674 [2.410 to 13.354] | 0.022 [0.014 to 0.034]
  III (At Delivery) | 2.518 [0.994 to 6.382] | 1.657 [0.602 to 4.561] | 6.152 [2.063 to 18.348] | 3.199 [1.138 to 8.994] | 2.591 [1.156 to 5.806] | 6.609 [2.877 to 15.182] | 0.023 [0.015 to 0.035]
  IV (Week 2) | 1.219 [0.577 to 2.573] | 0.831 [0.408 to 1.693] | 1.783 [0.883 to 3.599] | 1.912 [0.849 to 4.304] | 2.087 [1.187 to 3.671] | 1.700 [0.810 to 3.566] | 0.009 [0.007 to 0.013]
  IV (Month 1) | 1.198 [0.534 to 2.687] | 0.783 [0.369 to 1.661] | 1.563 [0.706 to 3.460] | 2.089 [1.004 to 4.347] | 1.219 [0.620 to 2.396] | 2.442 [1.444 to 4.128] | 0.013 [0.009 to 0.018]
  IV (At Delivery) | 1.690 [0.915 to 3.121] | 0.556 [0.250 to 1.235] | 1.624 [0.776 to 3.399] | 1.986 [0.893 to 4.416] | 1.821 [1.069 to 3.103] | 2.469 [1.457 to 4.182] | 0.012 [0.009 to 0.017]
  V (Week 2) | 0.114 [0.052 to 0.248] | 0.217 [0.080 to 0.587] | 0.522 [0.193 to 1.411] | 0.839 [0.286 to 2.466] | 0.755 [0.365 to 1.564] | 0.534 [0.204 to 1.397] | 0.014 [0.010 to 0.019]
  V (Month 1) | 0.115 [0.051 to 0.260] | 0.222 [0.074 to 0.663] | 0.610 [0.213 to 1.743] | 1.158 [0.435 to 3.083] | 0.750 [0.339 to 1.657] | 0.729 [0.293 to 1.817] | 0.014 [0.010 to 0.020]
  V (At Delivery) | 0.188 [0.098 to 0.360] | 0.252 [0.087 to 0.732] | 0.919 [0.344 to 2.458] | 1.462 [0.546 to 3.918] | 0.853 [0.413 to 1.759] | 0.901 [0.388 to 2.094] | 0.016 [0.011 to 0.023]

49. Secondary Outcome: GMCs of GBS Serotype-specific IgG at 2 Weeks, 1 Month After Vaccination and at Delivery: Maternal Participants Stage 3
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At 2 Weeks after Vaccination, 1 Month After Vaccination and at Delivery
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal)
Number analyzed (Participants) | 102 | 100
microgram per milliliter
  Ia (Week 2) | 9.233 [4.648 to 18.343] | 0.051 [0.027 to 0.096]
  Ia (Month 1) | 9.631 [5.178 to 17.914] | 0.054 [0.028 to 0.103]
  Ia (At Delivery) | 8.817 [4.969 to 15.643] | 0.052 [0.028 to 0.100]
  Ib (Week 2) | 0.815 [0.458 to 1.450] | 0.009 [0.006 to 0.013]
  Ib (Month 1) | 0.832 [0.465 to 1.488] | 0.011 [0.007 to 0.016]
  Ib (At Delivery) | 0.645 [0.377 to 1.103] | 0.011 [0.007 to 0.016]
  II (Week 2) | 40.234 [27.437 to 58.999] | 0.149 [0.103 to 0.216]
  II (Month 1) | 32.831 [21.455 to 50.240] | 0.140 [0.096 to 0.204]
  II (At Delivery) | 22.460 [14.817 to 34.043] | 0.146 [0.099 to 0.215]
  III (Week 2) | 6.422 [3.475 to 11.869] | 0.034 [0.023 to 0.050]
  III (Month 1) | 7.158 [4.141 to 12.375] | 0.034 [0.022 to 0.051]
  III (At Delivery) | 5.641 [3.486 to 9.129] | 0.031 [0.021 to 0.046]
  IV (Week 2) | 5.719 [3.952 to 8.275] | 0.014 [0.009 to 0.020]
  IV (Month 1) | 4.598 [3.229 to 6.549] | 0.014 [0.009 to 0.020]
  IV (At Delivery) | 2.708 [1.920 to 3.821] | 0.012 [0.009 to 0.018]
  V (Week 2) | 0.760 [0.427 to 1.352] | 0.013 [0.009 to 0.017]
  V (Month 1) | 0.732 [0.410 to 1.306] | 0.014 [0.010 to 0.020]
  V (At Delivery) | 0.452 [0.266 to 0.768] | 0.012 [0.009 to 0.017]

50. Secondary Outcome: GBS6 Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 1 Month After Vaccination and at Delivery: Maternal Participants Stage 2
Description: OPA for the 6 serotypes (Ia, Ib, II, III, IV, V) were determined in all participants for each blood sample.
Time Frame: At 1 Month After Vaccination and at Delivery
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal)
Number analyzed (Participants) | 39 | 39 | 28 | 26 | 39 | 40 | 103
Titer
  Ia (Month 1) | 13012.1 [8833.7 to 19166.7] | 7765.3 [4510.1 to 13369.8] | 14408.2 [8688.7 to 23892.6] | 9722.0 [5042.9 to 18742.6] | 8133.8 [3884.6 to 17031.1] | 23271.2 [16886.0 to 32070.9] | 200.2 [148.1 to 270.6]
  Ia (At delivery) | 10500.3 [5750.8 to 19172.5] | 7160.6 [4139.7 to 12386.1] | 7560.6 [4145.9 to 13788.0] | 10501.6 [5084.2 to 21691.3] | 11820.6 [6122.2 to 22822.9] | 13037.0 [8256.0 to 20586.8] | 228.0 [159.7 to 325.4]
  Ib (Month 1) | 11534.8 [6127.3 to 21714.3] | 10639.1 [5992.3 to 18889.3] | 9835.4 [4446.4 to 21755.7] | 9031.8 [3780.8 to 21575.3] | 13747.4 [7723.3 to 24470.3] | 20896.2 [12772.3 to 34187.4] | 864.9 [592.5 to 1262.5]
  Ib (At delivery) | 14876.0 [6608.3 to 33487.9] | 12259.3 [6958.6 to 21597.9] | 14665.8 [6990.4 to 30768.4] | 10741.1 [4206.8 to 27425.2] | 16005.8 [8790.7 to 29142.9] | 19050.4 [10640.3 to 34107.8] | 794.2 [512.8 to 1230.2]
  II (Month 1) | 9908.6 [6649.3 to 14765.6] | 5486.1 [3655.7 to 8232.9] | 16560.9 [9736.9 to 28167.2] | 8564.5 [4974.9 to 14744.2] | 9693.4 [6287.5 to 14944.5] | 22480.0 [14472.6 to 34917.9] | 856.3 [641.7 to 1142.6]
  II (At delivery) | 9573.5 [5948.3 to 15408.0] | 6521.0 [3963.2 to 10729.7] | 18640.8 [13002.6 to 26723.8] | 9305.9 [5201.3 to 16649.7] | 13197.3 [8444.8 to 20624.3] | 19559.7 [11908.5 to 32126.9] | 1012.0 [742.7 to 1378.8]
  III (Month 1) | 4026.7 [2234.9 to 7255.0] | 3285.5 [1802.0 to 5990.4] | 11207.9 [5496.5 to 22854.0] | 3884.7 [2298.0 to 6567.2] | 4829.8 [2615.6 to 8918.4] | 7463.5 [4309.8 to 12924.7] | 547.2 [398.6 to 751.2]
  III (At delivery) | 5105.3 [2701.9 to 9646.8] | 3959.5 [2200.6 to 7124.3] | 5229.1 [2638.7 to 10362.5] | 3850.2 [1890.0 to 7843.4] | 5669.2 [3175.7 to 10120.4] | 5209.2 [2752.3 to 9859.5] | 429.6 [300.8 to 5209.2]
  IV (Month 1) | 6591.5 [4596.8 to 9451.9] | 6087.6 [4249.5 to 8720.9] | 8773.7 [5381.7 to 14303.7] | 7862.5 [4642.8 to 13315.3] | 6576.7 [4303.1 to 10051.7] | 8570.4 [5776.1 to 12716.5] | 1303.1 [993.3 to 1709.4]
  IV (At delivery) | 8074.3 [5019.7 to 12987.6] | 6302.6 [4344.3 to 9143.7] | 7713.8 [5537.3 to 10745.9] | 7494.3 [4144.7 to 13551.0] | 7557.0 [5062.9 to 11279.9] | 7316.2 [4995.8 to 10714.5] | 1146.0 [851.4 to 1542.4]
  V (Month 1) | 3048.0 [2012.8 to 4615.7] | 5568.4 [3485.6 to 8896.0] | 7288.6 [3896.5 to 13633.6] | 5272.9 [2895.9 to 9600.9] | 4359.2 [2741.0 to 6932.6] | 5607.4 [3761.8 to 8358.4] | 790.8 [545.4 to 1146.6]
  V (At delivery) | 2450.4 [1564.1 to 3839.0] | 3109.0 [1777.9 to 5436.6] | 6309.7 [3524.3 to 11296.3] | 2145.3 [2145.3 to 7367.4] | 4642.9 [2857.4 to 7544.2] | 5364.8 [3361.9 to 8560.7] | 649.1 [443.5 to 949.9]

51. Secondary Outcome: GBS6 Serotype-Specific OPA Geometric Mean Titers (GMTs) at 1 Month After Vaccination and at Delivery: Maternal Participants Stage 3
Description: OPA for the 6 serotypes (Ia, Ib, II, III, IV, V) were determined in all participants for each blood sample.
Time Frame: At 1 Month After Vaccination and at Delivery
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Stage 3: GBS6 20 mcg Without AlPO4 (Infant): Infant participants born to the maternal participants were randomized to receive a single dose of 20 mcg of GBS6 vaccine without AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 102 | 100
Titer
  Ia: at 1 month | 11462.9 [7717.7 to 17025.6] | 196.1 [143.3 to 268.5]
  Ia: at delivery | 6228.2 [3987.0 to 9729.2] | 211.4 [146.0 to 306.0]
  Ib: at 1 month | 13306.1 [9230.1 to 19182.2] | 480.8 [316.5 to 730.3]
  Ib: at delivery | 7011.6 [4414.7 to 11136.1] | 481.6 [314.6 to 737.1]
  II: at 1 month | 35652.7 [27220.2 to 46697.5] | 1911.7 [1381.8 to 2644.6]
  II: at delivery | 22650.9 [16845.7 to 30456.6] | 1998.5 [1418.4 to 2816.0]
  III: at 1 month | 9064.7 [6412.0 to 12814.8] | 511.9 [362.8 to 722.3]
  III: at delivery | 5822.1 [3929.9 to 8625.3] | 561.7 [392.2 to 804.6]
  IV: at 1 month | 11800.6 [9297.8 to 14977.0] | 1152.1 [854.6 to 1553.2]
  IV: at delivery | 8242.0 [6327.8 to 10735.1] | 1164.0 [837.9 to 1617.0]
  V: at 1 month | 9258.1 [7138.7 to 12006.7] | 846.0 [569.0 to 1257.9]
  V: at delivery | 5501.3 [3875.7 to 7808.6] | 837.5 [530.6 to 1322.0]

52. Secondary Outcome: GMCs of GBS6 Serotype-Specific IgG Infant Participant at Birth: Infant Participants Stage 2
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At Birth
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 36 | 30 | 31 | 31 | 36 | 38 | 99
Microgram per milliliter
  Ia | 4.322 [1.291 to 14.471] | 10.978 [4.362 to 27.625] | 6.128 [0.996 to 37.710] | 11.089 [1.919 to 64.083] | 6.094 [1.435 to 25.870] | 22.159 [11.705 to 41.949] | 0.047 [0.025 to 0.091]
  Ib | 0.155 [0.034 to 0.712] | 0.182 [0.045 to 0.727] | 0.481 [0.056 to 4.113] | 0.427 [0.083 to 2.206] | 0.253 [0.084 to 0.766] | 0.655 [0.217 to 1.976] | 0.007 [0.005 to 0.011]
  II | 7.680 [2.851 to 20.690] | 1.935 [1.009 to 3.711] | 5.190 [1.314 to 20.507] | 4.522 [1.393 to 14.680] | 12.594 [4.814 to 32.948] | 16.979 [8.465 to 34.057] | 0.080 [0.054 to 0.117]
  III | 0.954 [0.219 to 4.148] | 1.009 [0.289 to 3.521] | 0.917 [0.118 to 7.109] | 0.906 [0.208 to 3.954] | 1.085 [0.302 to 3.902] | 3.417 [1.495 to 7.810] | 0.017 [0.011 to 0.026]
  IV | 0.993 [0.403 to 2.447] | 0.448 [0.165 to 1.215] | 0.759 [0.275 to 2.098] | 0.550 [0.193 to 1.564] | 1.104 [0.454 to 2.684] | 1.903 [1.033 to 3.505] | 0.007 [0.005 to 0.009]
  V | 0.084 [0.031 to 0.226] | 0.090 [0.025 to 0.327] | 0.183 [0.054 to 0.618] | 1.255 [0.267 to 5.908] | 0.327 [0.123 to 0.871] | 0.502 [0.199 to 1.267] | 0.010 [0.007 to 0.015]

53. Secondary Outcome: GMCs of GBS6 Serotype-Specific IgG Infant Participant at Birth: Infant Participants Stage 3
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At Birth
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 86 | 88
Microgram per milliliter
  Ia | 6.366 [3.343 to 12.122] | 0.048 [0.026 to 0.089]
  Ib | 0.466 [0.261 to 0.833] | 0.009 [0.006 to 0.014]
  II | 16.123 [10.030 to 25.916] | 0.134 [0.090 to 0.201]
  III | 3.609 [2.076 to 6.275] | 0.024 [0.016 to 0.036]
  IV | 2.124 [1.391 to 3.243] | 0.013 [0.009 to 0.020]
  V | 0.278 [0.160 to 0.481] | 0.011 [0.008 to 0.015]

54. Secondary Outcome: GBS6 Serotype-Specific OPA GMTs Measured at Birth: Infant Participants Stage 2
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At Birth
Population: Evaluable immunogenicity population.Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant)
Number analyzed (Participants) | 36 | 30 | 31 | 31 | 36 | 38 | 99
Titer
  Ia | 991.5 [428.9 to 2291.8] | 2116.3 [952.2 to 4703.4] | 1927.4 [792.8 to 4686.0] | 3053.1 [1203.9 to 7742.2] | 1459.1 [464.1 to 4587.1] | 7916.5 [4001.6 to 15661.4] | 91.3 [77.0 to 108.3]
  Ib | 410.3 [159.2 to 1057.5] | 357.2 [122.4 to 1042.1] | 986.5 [297.8 to 3268.6] | 1160.5 [411.1 to 3276.0] | 451.1 [190.9 to 1066.1] | 1879.2 [632.9 to 5579.7] | 137.1 [97.7 to 192.4]
  II | 440.3 [251.6 to 770.6] | 399.5 [212.8 to 750.0] | 689.0 [313.0 to 1516.8] | 606.8 [242.7 to 1517.1] | 1049.9 [440.7 to 2501.3] | 3262.2 [1355.4 to 7851.6] | 212.8 [186.2 to 243.3]
  III | 452.2 [203.9 to 1003.0] | 249.1 [119.0 to 521.4] | 698.4 [205.7 to 2371.5] | 479.0 [175.0 to 1311.3] | 634.2 [267.5 to 1503.2] | 766.9 [323.4 to 1818.7] | 79.2 [67.9 to 92.4]
  IV | 276.7 [174.6 to 438.4] | 379.3 [160.4 to 897.0] | 258.8 [170.3 to 393.2] | 439.2 [220.2 to 875.7] | 438.8 [195.6 to 984.5] | 1071.2 [484.0 to 2370.8] | 157.2 [122.8 to 201.3]
  V | 91.2 [67.3 to 123.8] | 162.4 [78.7 to 335.4] | 143.7 [71.5 to 289.1] | 521.2 [193.8 to 1401.3] | 219.1 [90.5 to 530.8] | 1189.4 [440.5 to 3211.4] | 98.3 [74.3 to 129.9]

55. Secondary Outcome: GBS6 Serotype-Specific OPA GMTs Measured at Birth: Infant Participants Stage 3
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: At Birth
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
Number analyzed (Participants) | 86 | 88
Titer
  Ia | 1173.7 [659.3 to 2089.1] | 89.5 [75.0 to 106.7]
  Ib | 1108.3 [590.7 to 2079.3] | 114.8 [90.1 to 146.3]
  II | 3639.4 [2310.4 to 5732.9] | 291.0 [219.3 to 386.1]
  III | 1005.6 [571.1 to 1770.5] | 77.1 [66.0 to 90.1]
  IV | 854.0 [550.4 to 1325.1] | 160.2 [128.7 to 199.4]
  V | 393.8 [227.6 to 681.3] | 127.8 [90.6 to 180.2]

ADVERSE EVENTS:
Time Frame: For Stage 1: From Day 1 up to 3.5 years post vaccination, For Stage 2 and 3: maximum up to 12 months post-delivery
Description: Same event may appear as non-SAE & SAE but are distinct events. Event may be serious in one participant & non-serious in another or one participant may have experienced both serious & non-serious events. Safety analysis set included all participants who received a primary dose of GBS6 vaccine or placebo.
Groups:
- Stage 2: GBS6 10 mcg With AlPO4 (Maternal): Maternal participants were randomized to receive a single dose of 10 μg of GBS6 vaccine with AlPO4, intramuscularly on Day 1.
Arm/Group | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1: Placebo (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) | Stage 1 Booster: Placebo (Nonpregnant) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 2: Placebo (Maternal) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) | Stage 2: Placebo (Infant) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) | Stage 3: Placebo (Maternal) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) | Stage 3: Placebo (Infant)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/11 | 0/7 | 0/8 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 1/120 | 0/40 | 1/39 | 0/40 | 0/40 | 0/40 | 0/40 | 2/118 | 0/108 | 0/108 | 3/104 | 2/105
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/11 | 0/7 | 0/8 | 7/40 | 18/40 | 9/40 | 11/40 | 8/40 | 14/40 | 30/120 | 17/40 | 19/39 | 15/40 | 12/40 | 19/40 | 14/40 | 60/118 | 21/108 | 23/108 | 45/104 | 46/105
Other Adverse Events (participants affected / at risk) | 17/22 | 17/22 | 18/22 | 9/11 | 7/7 | 8/8 | 30/40 | 36/40 | 31/40 | 27/40 | 34/40 | 36/40 | 98/120 | 27/40 | 19/39 | 22/40 | 26/40 | 20/40 | 21/40 | 66/118 | 91/108 | 90/108 | 78/104 | 81/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) (N=22) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) (N=22) | Stage 1: Placebo (Nonpregnant) (N=22) | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) (N=11) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) (N=7) | Stage 1 Booster: Placebo (Nonpregnant) (N=8) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: Placebo (Maternal) (N=120) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) (N=39) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) (N=40) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) (N=40) | Stage 2: Placebo (Infant) (N=118) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) (N=108) | Stage 3: Placebo (Maternal) (N=108) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) (N=104) | Stage 3: Placebo (Infant) (N=105)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound sepsis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Breech delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 3 | 9 | 4 | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 14 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accessory auricle (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Birth mark (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Cardiac malposition (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Congenital cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congenital hiatus hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 3 | 5 | 8 | 3 | 20 | 0 | 0 | 15 | 15
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 11 | 5 | 9 | 10 | 5 | 20 | 0 | 0 | 20 | 13
Gastrointestinal disorder congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 5
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 4
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 0 | 4 | 0 | 6 | 0 | 0 | 0 | 4
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 6 | 0 | 0 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia foetal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perinatal depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Factor VIII deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Preauricular cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Neonatal gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 9 | 0 | 9 | 9 | 9 | 9 | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenoviral conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neonatal bacterial pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neonatal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: GBS6 20 mcg With AlPO4 (Nonpregnant) (N=22) | Stage 1: GBS6 20 mcg Without AlPO4 (Nonpregnant) (N=22) | Stage 1: Placebo (Nonpregnant) (N=22) | Stage 1 Booster: GBS6 20 mcg With AlPO4 (Nonpregnant) (N=11) | Stage 1 Booster: GBS6 20 mcg Without AlPO4 (Nonpregnant) (N=7) | Stage 1 Booster: Placebo (Nonpregnant) (N=8) | Stage 2: GBS6 5 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 5 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: GBS6 10 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 10 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: GBS6 20 mcg With AlPO4 (Maternal) (N=40) | Stage 2: GBS6 20 mcg Without AlPO4 (Maternal) (N=40) | Stage 2: Placebo (Maternal) (N=120) | Stage 2: GBS6 5 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 5 mcg Without AlPO4 (Infant) (N=39) | Stage 2: GBS6 10 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 10 mcg Without AlPO4 (Infant) (N=40) | Stage 2: GBS6 20 mcg With AlPO4 (Infant) (N=40) | Stage 2: GBS6 20 mcg Without AlPO4 (Infant) (N=40) | Stage 2: Placebo (Infant) (N=118) | Stage 3: GBS6 20 mcg Without AlPO4 (Maternal) (N=108) | Stage 3: Placebo (Maternal) (N=108) | Stage 3: GBS6 20 mcg Without AlPO4 (Infant) (N=104) | Stage 3: Placebo (Infant) (N=105)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 2 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 4 | 2 | 4 | 2 | 0 | 2 | 2 | 7 | 4 | 9 | 3 | 4 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 12 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (NAUSEA/VOMITING) (Gastrointestinal disorders) | 2 | 3 | 7 | 1 | 1 | 5 | 6 | 3 | 8 | 6 | 6 | 9 | 32 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 30 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 8 | 7 | 10 | 4 | 1 | 5 | 15 | 18 | 15 | 15 | 19 | 17 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 44 | 0 | 0
Injection site discolouration (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (REDNESS) (General disorders) | 4 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (PAIN) (General disorders) | 9 | 8 | 7 | 9 | 3 | 4 | 15 | 6 | 16 | 6 | 19 | 14 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 19 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (SWELLING) (General disorders) | 3 | 2 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess bacterial (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 3 | 4 | 1 | 1 | 0 | 4
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 2 | 2 | 1 | 0 | 3 | 2 | 2 | 3 | 2 | 2 | 5 | 9 | 3 | 5 | 7 | 11 | 11 | 21 | 38 | 31 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 2 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 2 | 5 | 6 | 1 | 0 | 3 | 5 | 10 | 7 | 6 | 7 | 10 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 15 | 0 | 0
Headache (Nervous system disorders) | 1 | 5 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 9 | 9 | 12 | 5 | 2 | 6 | 12 | 19 | 12 | 13 | 13 | 16 | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 39 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 7 | 4 | 2 | 5 | 2 | 2 | 7 | 6 | 7 | 6 | 7
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 2 | 1 | 2 | 3 | 0 | 0 | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0
Sexually transmitted disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site rash (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 0 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amniotic fluid index decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2 | 2 | 1 | 2 | 4 | 4 | 1 | 5 | 6 | 8 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 14 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 10 | 7 | 6 | 7 | 10 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breech delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perinatal depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Breast engorgement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Vaginal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2 | 2 | 3 | 2 | 0 | 6 | 8 | 11 | 8 | 11
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suture insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inferior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Macrosomia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic haematoma obstetric (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida nappy rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 7 | 4 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 3 | 0 | 0 | 0 | 9 | 12 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 7 | 2 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 2 | 5 | 2 | 2 | 7 | 1 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 2 | 1 | 0 | 2 | 12 | 10 | 12 | 10
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 1 | 0 | 0 | 9 | 8 | 9 | 8
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bradycardia neonatal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tethered oral tissue (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinopathy of prematurity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 3 | 4 | 0 | 0 | 5 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 7
Conjunctivitis bacteria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obesity (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight gain poor (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Newborn head moulding (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cephalhaematoma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Jaundice neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0
Low birth weight baby (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Meconium stain (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premature baby (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0
Shoulder dystocia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 5 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 4 | 2
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Tachycardia foetal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema impetiginous (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurodevelopmental delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Episiotomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03765073/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT03765073/SAP_001.pdf